CLINICAL TRIAL: NCT03349671
Title: Second Trimester Doppler Indices and Placental Vascularity as Predictors of Intrauterine Growth Restriction
Brief Title: Predictors of Intrauterine Growth Restriction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: IUGRPET
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ultrasound — A 3D volume of the uterus will be acquired by transabdominal sonography. The sweep angle was set at 85º and the probe will be kept perpendicular to the placental plate. The placenta will be examined and the size of the volume box will be adapted in such a way that the placenta fitted into it completely. The volume will then stored for later offline analysis.

SUMMARY:
The main objectives of modern antenatal care programs are to identify high risk pregnancies then to predict any possibility of adverse pregnancy outcome as early as possible.

The earliest attempts to achieve this goal were possible with the introduction of ultrasound in obstetrical practice in the 1950s. A breakthrough that enabled obstetricians to directly visualize the fetus, placenta and amniotic fluid. At first 2-dimensional (2D) imaging was employed whereby fetal biometry and placental location were detected. Later on, Doppler measurements & 3-dimensional (3D) representation became feasible further revolutionizing this area

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female.
2. Pregnant ± 22 to 26 weeks gestation
3. Singleton pregnancy.
4. Consenting to participate

Exclusion Criteria:

1. Intrauterine fetal death
2. Diagnosed to have Any congenital anomalies
3. Symmetrical IUGR
4. Established fetal compromise that necessitates delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who meet the eligibility criteria of the study will be invited to participate and only those who will give agreement on the informed written consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The rate of preeclampsia during pregnancy. | 5 months
  number of women developed preeclampsia

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt